CLINICAL TRIAL: NCT06520644
Title: Effect of Interactive Training on Strength and Coordination in Cerebral Palsy
Brief Title: Effect Of Virtual Reality On Strength and Coordination in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shimaa Mohamed Reffat (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Shimaa Mohamed Reffat, lecturer of Physical Therapy Department for Pediatrics, Faculty of Physical Therapy, Cairo University, Egypt, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T. REC/012/003287
Record Dates: First submitted 2024-07-10; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial (RCT) as the selected children were divided randomly by sealed envelopes into two groups of equal number 15 children for each group. The investigator prepared 30 closed envelopes, with each envelope containing a card labeled as either group A or B. Each child legal guardian was asked to draw a closed envelope that determined whether he/she was allocated to Children in group A (control group N=15, Female =8, Male=7) received specially designed physical therapy program. Children in group B (study group=15, Female =10, Male=5) received the same program given to (group A) in addition to Wii-based interactive training. The sample size for this study was calculated using the G*power program 3.1.9 (G power program version 3.1, Heinrich-Heine-University, Düsseldorf, Germany) for one tailed test.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy program (Active Comparator): Children in group A (control group N=15, Female =8, Male=7)received specially designed physical therapy program.Facilitation of balance reactions from standing position including; standing on balance board, standing on one leg, weights shifting from standing position and stoops and recover from standing,Facilitation of counterpoising mechanism through instructing the child to kick ball from standing position as well as catching and throwing ball with his hands,Gait training activities including: walking on balance board, walking using different obstacles (rolls, wedges, stepper) and walking up and down stairs,Facilitation of protective reaction from standing position by pushing the child in different directions.Facilitation of rising mechanism through changing position e.g.: from lying to standing and from sitting to standing,Strengthening exercises for back and abdominal muscles as well as upper and lower limbs,Jumping in place and jumping a board.
  Interventions: Other: Traditional physical therapy program
- Traditional physical therapy program and Wii-based interactive training (Active Comparator): Children in group B (study group=15, Female =10, Male=5) received the same program given to (group A) in addition to Wii-based interactive training.Children in the study group received the same selected physical therapy program given to the control group in addition to 30 minutes Wii-based interactive training program. The frequency of the whole program will be three times per week, for three months.
  Nintendo Wii video game consists of console, remote, nunchuck and balance board. The Wii gaming system is based on wireless controller.The games used in this study include step basic, hula hoop, table tilt, jogging, jumping, single limb extension.
  Interventions: Device: Wii-based interactive training program; Other: Traditional physical therapy program

INTERVENTIONS:
Device: Wii-based interactive training program — include step basic, hula hoop, table tilt, jogging, jumping, single limb extension. Single limb extension
  Arms: Traditional physical therapy program and Wii-based interactive training
Other: Traditional physical therapy program — Facilitation of balance reactions from standing position including; standing on balance board, standing on one leg, weights shifting from standing position and stoops and recover from standing,Facilitation of counterpoising mechanism through instructing the child to kick ball from standing position as well as catching and throwing ball with his hands,Gait training activities including: walking on balance board, walking using different obstacles (rolls, wedges, stepper) and walking up and down stairs,Facilitation of protective reaction from standing position by pushing the child in different directions.Facilitation of rising mechanism through changing position e.g.: from lying to standing and from sitting to standing,Strengthening exercises for back and abdominal muscles as well as upper and lower limbs,Jumping in place and jumping a board.

SUMMARY:
ABSTRACT:

Purpose: To investigate the effect of interactive training on muscle strength and coordination in children with hemiparesis.

Materials and methods: This study involved 30 children of both sexes with unilateral cerebral palsy aged ranged 8 up to 10 years. A designed physical rehabilitation program was given to both groups. furthermore, study group received a wii fit virtual reality-based program. Muscle strength, bilateral coordination, running speed and agility were assessed by using Bruininks-Oseretsky test of motor proficiency, 2nd edition (BOT-2) while hip and knee extensor strength were assessed by lafayette hand-held dynamometer pre and post treatment program.

DETAILED DESCRIPTION:
INTRODUCTION Cerebral palsy (CP) is the most common disability of childhood that affects motor function because of injury to the developing brain . Cerebral Palsy is an umbrella term encompassing a heterogeneous group of permanent but not unchanging disorders of movement and posture that is caused by damage to the developing brain .

Children with CP show various motor impairments such as muscle weakness, spasticity, limited range of motion, and loss of selective motor function. These impairments make the development of normal gross motor function difficult. The focus of therapy in CP is to develop enough gross motor function for performing basic life activities independently . children with CP may experience a wide range of lifelong difficulties (such as cognitive impairment, epilepsy, communication difficulties, visual or hearing impairment, progressive musculoskeletal deformities, pain) .

Hemiplegia is a neurological disorder that is frequently detected in children with CP. It may provoke altered selective motor control, weakness, and spasticity. While one side is affected by the disorder, the contralateral side appears to maintain complete functionality. The consequent asymmetry has been proven to affect many daily-life tasks, such as walking .

Studies have proved that the gross motor skill disorder is an important factor hindering children with CP from participating in physical activities . Components of motor capabilities such as speed, agility, strength, coordination, balance, flexibility, durability are needed by CP. Speed and agility are essential components for the movement of CP. Speed is a qualified ability in addition to strength and endurance. Agility is a psychomotor skill that allows rapid change of movement direction without losing control and balance of movement.

The BOT-2 is norm-referenced, and it involves individually administered tasks with direct observation and assessment of a child in a structured environment. Evidence supporting the use of the BOT-2 to assess gross and fine motor proficiency of individuals aged 4 through 21. The BOT-2 had face validity of the items in that they reflect typical childhood motor activities also it had construct validation of the test . Lafayette manual muscle testing system is commonly used device that measure isometric lower limb muscle strength. Handheld dynamometer is used to assess lower limb strength. The test-retest interclass correlation coefficient ranged from 0.95 to 0.99 .

Virtual reality (VR) is a technology that provides a sense of presence in a real environment with the help of 3D pictures and animations formed in a computer environment and enable the person to interact with the objects in that environment . It was described as an improved form of human-computer interaction that allows the user to be part of and interact with a computer-generated environment . Virtual rehabilitation is a relatively new method in CP treatment that provides CP patients the opportunity to play an interactive game. In the recent years, there has been increasing interest in the use of the Nintendo Wii and Wii Fit (Wii) as virtual rehabilitation tools. This active video games system may allow children with CP to perform many types of activities they cannot do in the real world .

The Nintendo Wii FitTM, a computer game console, is an interesting example of a new exercise choice that could be used for improving strength, flexibility, fitness, postural stability, and general well-being of healthy adult and elderly . However, the main aim of the study to investigate the effect of interactive training on muscle strength and coordination in children with hemiparesis.

MATERIALS AND METHODS Design The study is a randomized controlled trial (RCT) as the selected children were divided randomly by sealed envelopes into two groups of equal number 15 children for each group. The investigator prepared 30 closed envelopes, with each envelope containing a card labeled as either group A or B. Each child legal guardian was asked to draw a closed envelope that determined whether he/she was allocated to Children in group A (control group N=15, Female =8, Male=7) received specially designed physical therapy program. Children in group B (study group=15, Female =10, Male=5) received the same program given to (group A) in addition to Wii-based interactive training. The sample size for this study was calculated using the G*power program 3.1.9 (G power program version 3.1, Heinrich-Heine-University, Düsseldorf, Germany) for one tailed test.

Participants Children with hemiparetic CP were recruited from the Outpatient Clinic of the Faculty of Physical Therapy, Cairo University. Thirty children were participating in the study 15 children in each group from both sexes aged 8 up to 10 years.

The study was approved by the Ethical Committee for Human Research at faculty of Physical therapy with reference number P.T. REC/012/003287.Participants legal guardian signed a written informed consent prior to participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-10 years old
* Children were included in the study had Mild degree of spasticity ranged from 1 to 1+ according to Modified Ashworth Scale[15].
* Motor skill level was at level I and II according to Gross Motor Function Classification System GMFCS[16].
* Able to follow instructions during evaluation and treatment

Exclusion Criteria:

* Children were excluded from the study had Cardiovascular or respiratory disorders.
* Botulinium muscular injection in the last 6 months.
* Surgical interference in lower limbs and/or spine.
* Muscloskeletal problems or fixed deformities in the spine and/or lower extremities.
* Seizures
* Visual or hearing impairment.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Bruininks-Oseretsky test of motor proficiency, 2nd edition (BOT-2) | through study completion, an average of 1 year
  The BOT-2 is norm-referenced, and it involves individually administered tasks with direct observation and assessment of a child in a structured environment. Evidence supporting the use of the BOT-2 to assess gross and fine motor proficiency of individuals aged 4 through 21[9]. The BOT-2 test consists of four composites and eight subtests including 53 items as follows: Fine manual control (fine motor precision, fine motor integration), Manual coordination (manual dexterity, upper limb coordination), Body Coordination (bilateral coordination, balance), Strength and Agility (running speed and agility, and strength
Lafayette manual muscle testing system | through study completion ,average of 1 year
  commonly used device that measure isometric lower limb muscle strength. Handheld dynamometer is used to assess lower limb strength. The test-retest interclass correlation coefficient ranged from 0.95 to 0.99

CONTACTS AND LOCATIONS:
Locations (1):
- Israa Ahmed Mohamed Shawki, Cairo, Egypt